CLINICAL TRIAL: NCT01283685
Title: Does Breathing Helium-Hyperoxia Increase the Tolerance of One-Legged Exercise in Ventilatory Limited Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Breathing Helium-Hyperoxia During Exercise in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSI-10q2109
Record Dates: First submitted 2010-07-06; First posted 2011-01-26 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise, Physical
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: breathing helium-hyperoxia — 40% O2, 60% He
Other: breathing supplemental oxygen — oxygen (4 L/min) provided by nasal cannula

SUMMARY:
Regular exercise can help patients with the lung disease, chronic obstructive pulmonary disease (COPD). But COPD patients have a hard time with training because of their breathing. To improve their program they can train with one leg at a time. Another way is to make their exercise easier by breathing helium. Putting two methods, one-legged and helium, together may improve their program even more. This project is planned to assess whether breathing helium improves their one-legged exercise endurance. If it does, then there may be a reason for combining one-legged exercise with breathing helium as part of their respiratory rehabilitation program. The aim of this study is to determine whether breathing helium-hyperoxia enables a further increase in the constant power endurance time during one-legged exercise in ventilatory limited subjects with COPD. The null hypothesis is that patients will have sufficient peripheral muscle limitation that ventilatory unloading using helium-hyperoxia will be of no additional benefit to exercise tolerance. The investigators hypothesize that patients with COPD are so ventilatory limited relative to their peripheral muscles that helium-hyperoxia will improve their exercise endurance.

DETAILED DESCRIPTION:
This is a randomized cross-over comparison trial determining the effects of helium-hyperoxia on the performance of muscle specific one-legged cycling. Each participant will complete two constant power exercise tests while cycling with their right leg only. The tests will be separated by at least 24 h. The conditions of the two tests will be the same except that, in randomized order, the participant will breathe helium-hyperoxia (40% O2, 60% He) through a mask, or room air unencumbered by a mask with supplemental oxygen (4 L/min) provided by nasal cannula.

Participants will perform three exercise tests. First they will complete one incremental power exercise test using both legs (exercise capacity) in a standardized manner. Then they will complete two constant power (exercise endurance) cycle ergometer tests to the limit of tolerance (symptom based); the intent is to set an exercise level that comparable to the ideal training session that a patient would experience in the respiratory rehabilitation program. The same exercise regimen will be used in these two sessions except that the participant will breathe helium-hyperoxia (40% O2, 60% He) in one session and room air, with supplemental oxygen (4 L/min) provided by nasal cannula, in the other. During all exercise sessions, heart rate, SaO2, and Borg scale ratings of dyspnoea and leg fatigue will be monitored. For each exercise test, participants will adhere to their usual medical regimens, not eat for 2 h before the test and not drink caffeinated beverages for 2 h before the test. All tests will be separated by at least 24 h.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD
* Cardiopulmonary impairment
* Ventilatory limitation

Exclusion Criteria:

* inability to communicate in English
* cardiac rhythm or circulatory compromise
* recent myocardial infarct
* moderate-severe aortic stenosis
* uncontrolled hypertension
* sustained cardiac arrhythmias
* untreated neoplasia
* lung surgery within the previous three months
* any other predominant co-morbidities, such as chronic heart failure, or treatments that might influence the results of exercise testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
tolerable duration of symptom-limited high-intensity exercise | 1 week

SECONDARY OUTCOMES:
heart rate | 1 week
oxygen saturation | 1 week
Breathlessness | 1 week
leg fatigue | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada